CLINICAL TRIAL: NCT02722057
Title: A Study in US Cystic Fibrosis Patients With the R117H-CFTR Mutation to Confirm the Long-term Safety and Effectiveness of Kalydeco, Including Patients <18 Years of Age, Combining Data Captured in the Cystic Fibrosis Foundation Registry From an Interventional Cohort and a Non-Interventional Cohort
Brief Title: A Study to Confirm the Long-term Safety and Effectiveness of Kalydeco in Patients With Cystic Fibrosis Who Have an R117H-CFTR Mutation, Including Pediatric Patients
Status: Completed | Type: Observational
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: VX15-770-122
Record Dates: First submitted 2016-03-22; First posted 2016-03-29 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

GROUPS / COHORTS (3):
- Cohort 1 - Interventional: The Interventional cohort will not be utilized.
- Cohort 2 - Non Interventional: A Non-Interventional Cohort comprising pediatric (<18 years of age) and adult R117H-CFTR patients treated with commercially-available Kalydeco.
- Cohort 3 - Historical: A Historical Cohort comprising data from an earlier time period for pediatric (<18 years of age) and adult patients with the R117H-CFTR mutation who have never been exposed to Kalydeco and matched on age, gender, and lung function to patients in the Non-Interventional Cohort.

SUMMARY:
The purpose of this study is to confirm the long-term safety and effectiveness of Kalydeco® (ivacaftor) in US CF patients with the R117H-CFTR mutation <18 years of age and to describe the long-term safety and effectiveness of Kalydeco in CF patients with the R117H-CFTR mutation overall and in patients ≥18 years. The long-term safety and effectiveness of Kalydeco will be examined in totality through the evaluation of the primary outcome measures.

DETAILED DESCRIPTION:
Patient follow-up (i.e., collection of outcomes data after treatment initiation) in the Non-Interventional Cohort will be at least 36 months. The study also includes retrieval of retrospective data entered into the registry for 36 months before the initiation of Kalydeco treatment, from patients matched for Non-Interventional Cohorts. This will permit a within-group comparison of outcomes before and after Kalydeco treatment for effectiveness and safety. The interventional cohort will not be utilized.

ELIGIBILITY:
Inclusion Criteria:

Non Interventional Cohort

* Male or female with confirmed diagnosis of CF
* Must have at least 1 allele of the R117H-CFTR mutation
* Enrolled in the US CFF Patient Registry
* With a record of Kalydeco treatment initiation from 01 January 2015 through 31 December 2016

Historical Cohort

* Patients with CF in the CFF Patient Registry as of 01 January 2009
* Must have at least 1 allele of the R117H-CFTR mutation
* Patients with no evidence of any prior Kalydeco exposure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Non Interventional Cohort - Patients Enrolled in the US CFF Patient Registry Historical Cohort - Patients with CF in the CFF Patient Registry as of 01 January 2009
Sampling Method: Non-Probability Sample
Enrollment: 368 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Lung function measurements (percent predicted forced expiratory volume in 1 second [FEV1] and forced vital capacity [FVC]) | 36 Months
  Spirometry will be performed according to the standard procedure at each site, and FEV1 values as recorded in the registry will be evaluated. All descriptive and summary data collected for FEV1 will be repeated for FVC
Pulmonary exacerbations, use of IV antibiotics | 36 Months
  Pulmonary exacerbation data will be collected as recorded in the registry.
Nutritional parameters (body mass index [BMI], BMI-for-age z-score, weight, and weight-for-age z-score) | 36 Months
  Height and weight measurements as recorded in the registry will be evaluated. BMI, BMI-for-age z-score, and weight-for-age z-score will be derived
Death or transplantation | 36 months
  Death will be collected from the registry database.
Hospitalizations | 36 Months
  Hospitalizations will be collected from the registry database.
Selected Complications (Symptomatic sinus disease, Pulmonary complications, CF-related diabetes (CFRD) and distal intestinal obstruction syndrome (DIOS), Hepatobiliary complications, Pancreatitis) | 36 Months
  Information for the above shown CF-related complications as recorded in the registry will be evaluated
Select pulmonary microorganisms (e.g., P. aeruginosa, S. aureus) | 36 Months
  Data on microorganisms as recorded in the registry will be evaluated